CLINICAL TRIAL: NCT03152825
Title: Stress Perfusion Cardiac Magnetic Resonance for Ischaemia and Viability Detection in Patients With Coronary Chronic Total Occlusions
Brief Title: Stress CMR in Patients With Coronary Chronic Total Occlusions
Acronym: CARISMA_CTO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Massimo Lombardi, Director of Multimodality Cardiac Imaging Unit, Ospedale San Donato
Other Study IDs: CARISMA_CTO
Record Dates: First submitted 2017-05-07; First posted 2017-05-15 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Coronary Chronic Total Occlusions
Keywords: myocardial ischaemia; myocardial viability; coronary chronic total occlusions; cardiac magnetic resonance; stress CMR
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Viable myocardium Group: At least ONE of the following:
  1. Late gadolinium enhancement <75%.
  2. Improvement in segmental function ≥1 grade during low dose dobutamine
  Interventions: Procedure: PCI
- Non-viable myocardium group: At least ONE of the following:
  1. Late gadolinium enhancement ≥75%.
  2. No improvement in segmental function during low dose dobutamine
  Interventions: Procedure: PCI
- Inducible ischaemia group: At least ONE of the following:
  * perfusion defect (≥ 1,5 segments) assessed during peak infusion of adenosine or dobutamine
  * new wall motion abnormalities or worsening ≥1 grade during peak infusion of dobutamine
  Interventions: Procedure: PCI
- Non-inducible ischaemia group: None of conditions qualifying for the "Inducible ischemia group"
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — percutaneous coronary intervention attempt

SUMMARY:
A total chronic occlusion (CTO) is defined as a coronary obstruction with TIMI 0 flow lasting at least 3 months.The prevalence of CTO in patients with coronary disease is about 10-40%. Coronary collateralizations may supply sufficient perfusion to retain tissue viability, but do not protect from myocardial ischaemia. In fact, percutaneous revascularization (PCI) of CTO lesions leads to improved symptoms, functional class, quality of life, higher left ventricular ejection fraction and improved survival in several observational studies. However, due to the higher rate of procedural complications and lower success rate of PCI than in other settings, it is attempted in only 10% of all CTO lesions. Myocardial viability/ischaemia assessment should be performed before PCI to avoid potential PCI-related complications and identify patients who might benefit most from myocardial revascularization, individualizing the risk-to-benefit ratio. In this regard, patients with stable coronary artery disease who have moderate-to-severe ischaemia are at higher risk of event rates (death or MI of ~5%/year) and plausibly represent the best target for PCI.

Cardiac MRI (CMR) provide a reliable assessment of both myocardial ischaemia and viability. Using late gadolinium enhancement (LGE) sequences, myocardial segments with LGE >75% of transmurality do not show any improvement in contractility even after revascularization, representing a subset of patients in which CTO PCI may be futile. Viability assessment by CMR may be also performed with low dose dobutamine infusion; in patients with CTO and akinetic segments, contractility improvement at low dose dobutamine may predict functional recovery in the follow-up. Myocardial ischaemia may be assessed by CMR with high accuracy, identifying perfusion defects during pharmacological-induced hyperemia and/or regional wall motion abnormalities during inotrope infusion.

This study is designed to verify the hypothesis that myocardial ischaemia and viability assessed by CMR could identify patients who are more likely to benefit from PCI in terms of improvement in left ventricular remodeling, functional recovery and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Angiographic diagnosis of Coronary Chronic Total Occlusion (TIMI 0 lasting more than 3 months, if known)
* baseline stress CMR
* signed informed consent

Exclusion Criteria:

* CMR contraindications
* severe CKD
* contraindications to adenosine or dobutamine
* unable/unwilling to sign informed consent
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with angiographic evidence of CTO with planned PCI.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Left ventricular mechanical improvement after PCI | 12 +/- 3 months
  At least ONE of the following:
  * Delta ejection fraction ≥ 5%
  * Segmental function improvement ≥1 grade
  * Delta end-diastolic volume ≥ 10%
  * Delta end-systolic volume ≥ 10%

SECONDARY OUTCOMES:
Stress ischaemia improvement after PCI | 12 +/- 3 months
  At least ONE of the following stress CMR (adenosine or dobutamine) findings:
  _<1.5 segments perfusion defect
  _≥1 grade improvement in segmental wall motion abnormalities
Quality of life assessed by Seattle Angina Questionnaire (SAQ) | 12+/-3 months
  Delta SAQ score
Major cardiovascular events | 12+/- 3 months
  all-cause death, death for cardiovascular cause, life-threatening arrythmia, hospitalization for heart failure, myocardial infarction, target vessel revascularization

OTHER OUTCOMES:
CMR to identify re-occlusion of CTO | 12 +/- 3 months
  Correlate angiographic CTO re-occlusion and/or critical re-stenosis with at least ONE of the following stress CMR parameters:
  * Segmental perfusion defect ≥1.5
  * New segmental contractility impairment
  * Delta ejection fraction, end-diastolic,end-systolic volume

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Lombardi, MD, Principal Investigator — Policlinico San Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

REFERENCES:
- [Background] Stone GW, Kandzari DE, Mehran R, Colombo A, Schwartz RS, Bailey S, Moussa I, Teirstein PS, Dangas G, Baim DS, Selmon M, Strauss BH, Tamai H, Suzuki T, Mitsudo K, Katoh O, Cox DA, Hoye A, Mintz GS, Grube E, Cannon LA, Reifart NJ, Reisman M, Abizaid A, Moses JW, Leon MB, Serruys PW. Percutaneous recanalization of chronically occluded coronary arteries: a consensus document: part I. Circulation. 2005 Oct 11;112(15):2364-72. doi: 10.1161/CIRCULATIONAHA.104.481283. No abstract available. PMID 16216980
- [Background] Shah PB. Management of coronary chronic total occlusion. Circulation. 2011 Apr 26;123(16):1780-4. doi: 10.1161/CIRCULATIONAHA.110.972802. No abstract available. PMID 21518991
- [Background] Baim DS, Kwong RY. Is magnetic resonance image guidance the key to opening chronic total occlusions? Circulation. 2006 Feb 28;113(8):1053-5. doi: 10.1161/CIRCULATIONAHA.105.609263. No abstract available. PMID 16505189
- [Background] Kahn JK. Angiographic suitability for catheter revascularization of total coronary occlusions in patients from a community hospital setting. Am Heart J. 1993 Sep;126(3 Pt 1):561-4. doi: 10.1016/0002-8703(93)90404-w. PMID 8362709
- [Background] Christofferson RD, Lehmann KG, Martin GV, Every N, Caldwell JH, Kapadia SR. Effect of chronic total coronary occlusion on treatment strategy. Am J Cardiol. 2005 May 1;95(9):1088-91. doi: 10.1016/j.amjcard.2004.12.065. PMID 15842978
- [Background] Grantham JA, Jones PG, Cannon L, Spertus JA. Quantifying the early health status benefits of successful chronic total occlusion recanalization: Results from the FlowCardia's Approach to Chronic Total Occlusion Recanalization (FACTOR) Trial. Circ Cardiovasc Qual Outcomes. 2010 May;3(3):284-90. doi: 10.1161/CIRCOUTCOMES.108.825760. Epub 2010 Apr 13. PMID 20388873
- [Background] Cheng AS, Selvanayagam JB, Jerosch-Herold M, van Gaal WJ, Karamitsos TD, Neubauer S, Banning AP. Percutaneous treatment of chronic total coronary occlusions improves regional hyperemic myocardial blood flow and contractility: insights from quantitative cardiovascular magnetic resonance imaging. JACC Cardiovasc Interv. 2008 Feb;1(1):44-53. doi: 10.1016/j.jcin.2007.11.003. PMID 19393143
- [Background] Pujadas S, Martin V, Rossello X, Carreras F, Barros A, Leta R, Alomar X, Cinca J, Sabate M, Pons-Llado G. Improvement of myocardial function and perfusion after successful percutaneous revascularization in patients with chronic total coronary occlusion. Int J Cardiol. 2013 Oct 30;169(2):147-52. doi: 10.1016/j.ijcard.2013.08.017. Epub 2013 Aug 15. PMID 24120215
- [Background] Christakopoulos GE, Christopoulos G, Carlino M, Jeroudi OM, Roesle M, Rangan BV, Abdullah S, Grodin J, Kumbhani DJ, Vo M, Luna M, Alaswad K, Karmpaliotis D, Rinfret S, Garcia S, Banerjee S, Brilakis ES. Meta-analysis of clinical outcomes of patients who underwent percutaneous coronary interventions for chronic total occlusions. Am J Cardiol. 2015 May 15;115(10):1367-75. doi: 10.1016/j.amjcard.2015.02.038. Epub 2015 Feb 18. PMID 25784515
- [Background] Hoebers LP, Claessen BE, Elias J, Dangas GD, Mehran R, Henriques JP. Meta-analysis on the impact of percutaneous coronary intervention of chronic total occlusions on left ventricular function and clinical outcome. Int J Cardiol. 2015;187:90-6. doi: 10.1016/j.ijcard.2015.03.164. Epub 2015 Mar 17. PMID 25828320
- [Background] Jang WJ, Yang JH, Choi SH, Song YB, Hahn JY, Choi JH, Kim WS, Lee YT, Gwon HC. Long-term survival benefit of revascularization compared with medical therapy in patients with coronary chronic total occlusion and well-developed collateral circulation. JACC Cardiovasc Interv. 2015 Feb;8(2):271-279. doi: 10.1016/j.jcin.2014.10.010. PMID 25700750
- [Background] Valenti R, Migliorini A, Signorini U, Vergara R, Parodi G, Carrabba N, Cerisano G, Antoniucci D. Impact of complete revascularization with percutaneous coronary intervention on survival in patients with at least one chronic total occlusion. Eur Heart J. 2008 Oct;29(19):2336-42. doi: 10.1093/eurheartj/ehn357. Epub 2008 Aug 5. PMID 18682446
- [Background] Kim RJ, Wu E, Rafael A, Chen EL, Parker MA, Simonetti O, Klocke FJ, Bonow RO, Judd RM. The use of contrast-enhanced magnetic resonance imaging to identify reversible myocardial dysfunction. N Engl J Med. 2000 Nov 16;343(20):1445-53. doi: 10.1056/NEJM200011163432003. PMID 11078769
- [Background] Selvanayagam JB, Kardos A, Francis JM, Wiesmann F, Petersen SE, Taggart DP, Neubauer S. Value of delayed-enhancement cardiovascular magnetic resonance imaging in predicting myocardial viability after surgical revascularization. Circulation. 2004 Sep 21;110(12):1535-41. doi: 10.1161/01.CIR.0000142045.22628.74. Epub 2004 Sep 7. PMID 15353496
- [Background] Wagner A, Mahrholdt H, Holly TA, Elliott MD, Regenfus M, Parker M, Klocke FJ, Bonow RO, Kim RJ, Judd RM. Contrast-enhanced MRI and routine single photon emission computed tomography (SPECT) perfusion imaging for detection of subendocardial myocardial infarcts: an imaging study. Lancet. 2003 Feb 1;361(9355):374-9. doi: 10.1016/S0140-6736(03)12389-6. PMID 12573373
- [Background] Baks T, van Geuns RJ, Duncker DJ, Cademartiri F, Mollet NR, Krestin GP, Serruys PW, de Feyter PJ. Prediction of left ventricular function after drug-eluting stent implantation for chronic total coronary occlusions. J Am Coll Cardiol. 2006 Feb 21;47(4):721-5. doi: 10.1016/j.jacc.2005.10.042. Epub 2006 Jan 26. PMID 16487835
- [Background] Kirschbaum SW, Baks T, van den Ent M, Sianos G, Krestin GP, Serruys PW, de Feyter PJ, van Geuns RJ. Evaluation of left ventricular function three years after percutaneous recanalization of chronic total coronary occlusions. Am J Cardiol. 2008 Jan 15;101(2):179-85. doi: 10.1016/j.amjcard.2007.07.060. Epub 2007 Dec 3. PMID 18178403
- [Background] Wellnhofer E, Olariu A, Klein C, Grafe M, Wahl A, Fleck E, Nagel E. Magnetic resonance low-dose dobutamine test is superior to SCAR quantification for the prediction of functional recovery. Circulation. 2004 May 11;109(18):2172-4. doi: 10.1161/01.CIR.0000128862.34201.74. Epub 2004 Apr 26. PMID 15117834
- [Background] Bellenger NG, Yousef Z, Rajappan K, Marber MS, Pennell DJ. Infarct zone viability influences ventricular remodelling after late recanalisation of an occluded infarct related artery. Heart. 2005 Apr;91(4):478-83. doi: 10.1136/hrt.2004.034918. PMID 15772205
- [Background] Fiocchi F, Sgura F, Di Girolamo A, Ligabue G, Ferraresi S, Rossi R, D'Amico R, Modena MG, Torricelli P. Chronic total coronary occlusion in patients with intermediate viability: value of low-dose dobutamine and contrast-enhanced 3-T MRI in predicting functional recovery in patients undergoing percutaneous revascularisation with drug-eluting stent. Radiol Med. 2009 Aug;114(5):692-704. doi: 10.1007/s11547-009-0426-2. Epub 2009 Jun 23. English, Italian. PMID 19551341
- [Background] Schwitter J, Arai AE. Assessment of cardiac ischaemia and viability: role of cardiovascular magnetic resonance. Eur Heart J. 2011 Apr;32(7):799-809. doi: 10.1093/eurheartj/ehq481. Epub 2011 Mar 11. PMID 21398645
- [Background] Jahnke C, Nagel E, Gebker R, Kokocinski T, Kelle S, Manka R, Fleck E, Paetsch I. Prognostic value of cardiac magnetic resonance stress tests: adenosine stress perfusion and dobutamine stress wall motion imaging. Circulation. 2007 Apr 3;115(13):1769-76. doi: 10.1161/CIRCULATIONAHA.106.652016. Epub 2007 Mar 12. PMID 17353441
- [Background] Gebker R, Jahnke C, Manka R, Hamdan A, Schnackenburg B, Fleck E, Paetsch I. Additional value of myocardial perfusion imaging during dobutamine stress magnetic resonance for the assessment of coronary artery disease. Circ Cardiovasc Imaging. 2008 Sep;1(2):122-30. doi: 10.1161/CIRCIMAGING.108.779108. Epub 2008 Jul 30. PMID 19808529
- [Background] Gebker R, Frick M, Jahnke C, Berger A, Schneeweis C, Manka R, Kelle S, Klein C, Schnackenburg B, Fleck E, Paetsch I. Value of additional myocardial perfusion imaging during dobutamine stress magnetic resonance for the assessment of intermediate coronary artery disease. Int J Cardiovasc Imaging. 2012 Jan;28(1):89-97. doi: 10.1007/s10554-010-9764-3. Epub 2010 Dec 14. PMID 21153708